CLINICAL TRIAL: NCT00526162
Title: Clinical Study to Evaluate System Safety and Clinical Performance of the ConsultaTM CRT-D Device
Brief Title: ConsultaTM CRT-D Clinical Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2019-03

CONDITIONS: Tachyarrhythmias; Heart Failure; Ventricular Dysfunction
MeSH Terms: conditions — Tachycardia; Heart Failure; Ventricular Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implantation of Consulta CRT-D (Experimental): Patients have an implant attempt with a Bi-ventricular Implantable Cardioverter Defibrillator
  Interventions: Device: Bi-ventricular Implantable Cardioverter Defibrillator

INTERVENTIONS:
Device: Bi-ventricular Implantable Cardioverter Defibrillator — Implantation of a Bi-ventricular Implantable Cardioverter Defibrillator
  Other Names: ConsultaTM

SUMMARY:
The purpose of the Consulta clinical study is to evaluate the overall system safety and clinical performance of the Consulta Implantable Cardioverter Defibrillator with Cardiac Resynchronization Therapy (CRT-D).

DETAILED DESCRIPTION:
The Consulta CRT-D is an investigational bi-ventricular device that provides atrial and ventricular tachyarrhythmia detection and therapy, cardioversion, defibrillation and cardiac resynchronization therapy.

The study will be a prospective, non-randomized, multicenter clinical study, conducted in approximately 18 centers.

To allow for sufficient experience with the device, a maximum of 80 subjects may be implanted with the Consulta device. Data will be collected at baseline (enrollment), implant, 1-, 3-, and 6- months post implant and every 6 months thereafter or until study closure (whichever occurs first), unscheduled follow-up visits, System Modifications, Technical Observations, Study Deviations, Study Exit, upon notification of new or updated Adverse Events and in case of death.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an indication for a defibrillator.
* Patients who are optimally treated with medication.
* Patients who are New York Heart Association (NYHA) Class III or IV

Exclusion Criteria:

* Patients with a life expectancy less than the duration of the study.
* Patients with medical conditions that preclude the testing required for all patients by the study protocol or that otherwise limit study participation required for all patients.
* Patients with mechanical tricuspid heart valves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Consulta Clinical Study Team, Study Chair — Medtronic Cardiac Rhythm and Heart Failure
Locations (1):
- Hospital, Bonn, Germany

REFERENCES:
- [Derived] Murgatroyd FD, Helmling E, Lemke B, Eber B, Mewis C, van der Meer-Hensgens J, Chang Y, Khalameizer V, Katz A. Manual vs. automatic capture management in implantable cardioverter defibrillators and cardiac resynchronization therapy defibrillators. Europace. 2010 Jun;12(6):811-6. doi: 10.1093/europace/euq053. Epub 2010 Mar 14. PMID 20231152

RESULTS

PARTICIPANT FLOW:
Groups:
- Consulta Implant: Patients implanted with a Consulta device
Period: Overall Study
Arm/Group | Consulta Implant
Started | 83
Completed | 80
Not Completed | 3
Not completed — Device not implanted | 3

BASELINE CHARACTERISTICS:
Groups:
- Consulta Implant: Patients implanted with a Consulta Cardiac Resynchronization Therapy (CRT)-D device
Arm/Group | Consulta Implant
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 62
Region of Enrollment [Number; unit: participants]
  Germany | 23
  Israel | 15
  United Kingdom | 11
  Netherlands | 7
  Norway | 6
  Denmark | 5
  Switzerland | 5
  Austria | 4
  France | 3
  Sweden | 2

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Unanticipated Serious Adverse Device Effects at 1-month Post Implant.
Description: Percentage of subjects without an unanticipated serious adverse device effects at 1-month post implant.Only subjects implanted with a Consulta device that were followed at least 28 days post-implant or have had a unanticipated device effect within 28 days after implant were included in the analysis.
Time Frame: 1 month
Population: Only subjects implanted with a Consulta device that were followed at least 28 days post-implant or have had a unanticipated device effect within 28 days after implant were included in the analysis.
Measure: Number (97.5% Confidence Interval); unit: percentage of patients
Arm/Group | Consulta Implant
Number analyzed (Participants) | 80
percentage of patients | 100 [90 to 100]
Statistical Analysis 1: Comparison: Consulta Implant; Test type: Other; p < 0.03, One proportion binomial exact — Using a confidence interval of 97%, the exact binomial upper confidence bound was 9.5% which is lower than the 10% set for the primary safety objective. Therefore, the actual p-value has not been calculated further; percentage = 0 — The confidence interval was calculated based on 35 patients who completed 1-month follow-up at interim analysis

2. Secondary Outcome: Adverse Events
Description: Number of Adverse Events reported in the implanted subjects.
Time Frame: 1 month
Measure: Number; unit: number of adverse events
Groups:
- Consulta Implant: Patients with a Consulta device implanted
Arm/Group | Consulta Implant
Number analyzed (Participants) | 80
number of adverse events | 70

3. Secondary Outcome: System Performance Assessed by Holter Records
Description: The first 20 digital Holter records that were successfully collected in the total of 80 implanted subjects were analysed on observation of device features, ventricular arrhythmia detection times and device classification of ventricular arrhythmias.
Time Frame: 1 month follow-up
Measure: Number; unit: number of Holter recordings
Groups:
- Consulta Implant: The first 20 patients implanted with a Consulta device that has a successful Holter recording
Arm/Group | Consulta Implant
Number analyzed (Participants) | 20
number of Holter recordings | 20

4. Secondary Outcome: System Performance Assessed by Save to Disk Files
Description: 94 Save to Disk files were reviewed on observation of device features, ventricular arrhythmia detection times and device classification of ventricular arrhythmias.
Time Frame: 1 month follow-up
Measure: Number; unit: number of Save to Disk files
Groups:
- Implantation of Consulta CRT-D: Patients implanted with a Bi-ventricular Implantable Cardioverter Defibrillator
Arm/Group | Implantation of Consulta CRT-D
Number analyzed (Participants) | 80
number of Save to Disk files | 94

5. Secondary Outcome: System Performance Assessed by Technical Observations
Description: Reported technical observations will be reviewed to determine if there are any device performance issues.
Time Frame: 1 month follow-up
Measure: Number; unit: number of Technical Observations
Groups:
- Implantation of Consulta CRT-D: Patients that are successfully implanted with a Bi-ventricular Implantable Cardioverter Defibrillator
Arm/Group | Implantation of Consulta CRT-D
Number analyzed (Participants) | 80
number of Technical Observations | 3

ADVERSE EVENTS:
Time Frame: From implant to 1 month follow-up visit
Groups:
- Consulta Implant: Patients implanted with a Consulta CRT-D device
Arm/Group | Consulta Implant
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 18/80
Other Adverse Events (participants affected / at risk) | 33/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Consulta Implant (N=80)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atypical Angina (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Cardiac Perforation (Surgical and medical procedures) | 1 (1)
Cardiac Failure (Cardiac disorders) | 2 (4)
Epistaxis (Injury, poisoning and procedural complications) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Implant site Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Lead dislodgement (Injury, poisoning and procedural complications) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 3 (3)
Perineal abscess (Congenital, familial and genetic disorders) | 1 (1)
Renal Failure (Injury, poisoning and procedural complications) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1)
Suicide (Social circumstances) | 1 (1)
Ventricular fibrillation (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Consulta Implant (N=80)
Amaurosis Fugax (Eye disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Increased blood glucose (Metabolism and nutrition disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Coronary sinus dissection (Injury, poisoning and procedural complications) | 1 (1)
Device malfunction (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac Failure (Cardiac disorders) | 5 (5)
Elevated pacing thresholds (Injury, poisoning and procedural complications) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Implant site haematoma (Injury, poisoning and procedural complications) | 2 (2)
Herpes Zoster (Renal and urinary disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Implant site pain (Injury, poisoning and procedural complications) | 2 (2)
Inappropriate device programming (Injury, poisoning and procedural complications) | 2 (2)
Phrenic nerve stimulation (Injury, poisoning and procedural complications) | 3 (3)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain (Gastrointestinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators to publish study results per the publication plan/protocol following Medtronic's review to determine whether Confidential Information (CI) is disclosed. Any such CI is deleted prior to publication/presentation. Medtronic may not censor/interfere with the publication except as described. Investigators may not publish any single-site publications until the main multi-site study publication has occurred.